CLINICAL TRIAL: NCT05807100
Title: Analyzing the Relationship Between Periodontal Health Status and Alzheimer's Disease
Brief Title: Investigation of Alzheimer's Disease and Periodontal Status
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: KKARADURAN001
Record Dates: First submitted 2023-03-13; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease; Periodontal Diseases
Keywords: Alzheimer's Disease; Cognitive Decline; Periodontal Disease; Periodontitis; Occlusion; Chewing
MeSH Terms: conditions — Alzheimer Disease; Periodontal Diseases; Cognitive Dysfunction; Periodontitis; Bites and Stings

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stage I: Stage I Alzheimer's Group (n=42): Individuals diagnosed with probable Alzheimer's disease with mild (early stage) dementia according to the Clinical Dementia Rating Scale.
  Interventions: Diagnostic Test: Baseline Standardized Mini Mental Test; Diagnostic Test: 6th month Standardized Mini Mental Test
- Stage II: Stage II Alzheimer's Group (n=29): Individuals diagnosed with probable Alzheimer's disease with moderate (moderate stage) dementia according to the Clinical Dementia Rating Scale.
  Interventions: Diagnostic Test: Baseline Standardized Mini Mental Test; Diagnostic Test: 6th month Standardized Mini Mental Test
- Stage III: Stage III Alzheimer's Group (n=19): Individuals diagnosed with probable Alzheimer's disease with severe (advanced stage) dementia according to the Clinical Dementia Rating Scale.
  Interventions: Diagnostic Test: Baseline Standardized Mini Mental Test; Diagnostic Test: 6th month Standardized Mini Mental Test

INTERVENTIONS:
Diagnostic Test: Baseline Standardized Mini Mental Test — Cognitive status assessment was done with Standardized Mini Mental Test.
Diagnostic Test: 6th month Standardized Mini Mental Test — Cognitive status assessment was done with Standardized Mini Mental Test.
  Other Names: Periodontal Examination: Toothed/edentulous condition, occlusal relationship type and periodontal status were evaluated by periodontal examination.

SUMMARY:
The aim of this study is to investigate the effect of the current periodontal status on the progression rate of AD.

DETAILED DESCRIPTION:
Although much is known about its pathogenesis, Alzheimer's disease (AD) is still a terminal disease. For this reason, the correct evaluation and treatment of the risk factors of the disease gains importance in the prevention of the disease. Chronic inflammation, such as periodontal disease, can speed up the onset and progression of AD. The study aimed to investigate the relationship between periodontal status and the rate of progression of dementia in individuals diagnosed with Alzheimer's disease.

In this study, 90 individuals with AD, who were classified as Stage I, Stage II, and Stage III according to the Clinical Dementia Rating Scale. Baseline and 6th month cognitive status assessments of participants who met the inclusion criteria were performed in the Department of Neurology using SMMT. At the 6th month control appointment in the Neurology Department, the participants were referred to the Periodontology Department for oral examinations.

In the Periodontology Department, dental anamnesis of the patients was taken and intraoral examinations were performed. Periodontal examination of all existing teeth of all participants with at least one remaining tooth (excluding third molars) with a Williams-marked periodontal probe (Hu-Friedy, Chicago, Illinois, USA) and all molars and maxillary first premolars with Nabers probe (PQ2N, Hu-Friedy, Chicago, Illinois, USA) was performed and records %P (plak percentage), %BOP (percentage bleeding on probing), CAL (clinical attachment level), PPD (probing pocket depth). The position of the gingival margin and PPD were measured at six sites/teeth (including/excluding third molars). The CAL was then calculated from these measurements. In 2017, periodontal status was determined according to the decisions of the World Workshop on Periodontal and Peri-implant Diseases and Classification of Conditions. The current occlusal relationship status of all patients was evaluated using the Eichner Index and classified as Type 1 (A1-A2-A3-B1) , Type 2 (B2-B3) and Type 3 (B4-C1-C2-C3).

ELIGIBILITY:
Inclusion Criteria:

* Those who have been diagnosed with probable Alzheimer's disease in the age range of 50-89
* Do not have dementia other than Alzheimer type dementia.
* Does not have a psychiatric disorder effecting cognitive status and does not use drugs that effect cognitive status.
* Those who have other existing systemic diseases (cardiovascular disease, diabetes) under control other than Alzheimer's disease.
* Not using regular anti-inflammatory and corticosteroids
* C-Reactive Protein (CRP) value was measured within 6 months prior to the date of inclusion in the study.
* Non-smoker and no alcohol intake
* Have not received any dental treatment in the last 1 year
* In those with less than 10 teeth, the edentulousness was prosthetically rehabilitated.

Exclusion Criteria:

-

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with mild/moderate/severe probable Alzheimer's disease according to the Clinical Dementia Rating Scale who meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Change in Standardized Mini Mental Test (SMMT) score at 6 months | Baseline and 6th month
  The baseline SMMT score was recorded. After 6 months, the 6th month SMMT score was recorded. Change in SMMT score at 6 months= Baseline SMMT score-6th SMMT score.

SECONDARY OUTCOMES:
Alzheimer's disease stage | Baseline
  The stage of Alzheimer's disease was determined according to the clinical dementia rating scale.
  Stage I: Mild, Stage II: Moderate, Stage III: Severe.
Gender | Baseline
  The gender distribution of Alzheimer's patients was divided into male and female.
Age | Baseline
  Ages of Alzheimer's patients were determined.
Number of Alzheimer's patient with systemic disease | Baseline
  The current systemic conditions of Alzheimer's patients were evaluated and those with diabetes mellitus and cardiovascular disease were determined.
Presence of periodontal disease | 6th month
  Alzheimer patients were evaluated according to the presence and absence of active periodontal disease.
Plaque percentage (%P) | 6th month
  It is an index that shows the amount of microbial dental plaque on the teeth.
Bleeding on probing percentage (%BOP) | 6th month
  Bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus.
Periodontal probing depth (PPD) (mm) | 6th month
  The distance from the gingival margin to pocket base.
Clinical attachment level (CAL) (mm) | 6th month
  The clinical attachment level is the distance between the enamel-cementum junction and the gingival sulcus.
Number of teeth | 6th month
  The number of teeth present in Alzheimer's patients was determined.
Occlusal relationship type | 6th month
  Alzheimer's patients were classified according to the Eichner Index (A1-A2-A3-B1-B2-B3-B4-C1-C2-C3). They were evaluated according to their occlusal relationship status and classified as Type 1, Type 2 and Type 3.
  * Type 1: A1-A2-A3-B1
  * Type 2: B2-B3
  * Type 3: B4-C1-C2-C3
C-Reactive Protein (CRP) (mg/l) | between baseline and -6th month
  C-Reactive Protein (CRP) is a protein found in blood plasma whose circulating concentration is associated with inflammation.
Neutrophil ratio (NEUT%) | between baseline and -6th month
  It refers to the percentage of circulating neutrophils to total white blood cells.
Lymphocyte ratio (LYMPH%) | between baseline and -6th month
  It refers to the percentage of circulating lymphocytes to total white blood cells.
Neutrophil count (10*3/uL) | between baseline and -6th month
  It is demonstrates the number of neutrophils in the peripheral blood.
Lymphocyte count (10*3/uL) | between baseline and -6th month
  It is demonstrates the number of lymphocytes in the peripheral blood.
Neutrophil-to-lymphocyte ratio (NLR) | between baseline and -6th month
  Neutrophil-to-lymphocyte ratio (NLR) is calculated by dividing the absolute number of neutrophils by absolute number of lymphocytes.
Mean platelet volume (fL) (MPV) | between baseline and -6th month
  Mean platelet volume (MPW) is a measure of the average size of the platelets.
Platelet distribution width (fL) (PDW) | between baseline and -6th month
  Platelet distribution width (PDW) reflects the variability in platelet size distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet AYDOĞDU, Study Director — Bezmialem Vakif University; Özlem GELİŞİN, Study Chair — Bezmialem Vakif University; Şadiye GÜNPINAR, Study Chair — Bezmialem Vakif University; Kübra KARADURAN, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih/Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared if requested.

REFERENCES:
- [Derived] Karaduran K, Aydogdu A, Gelisin O, Gunpinar S. Investigating the potential clinical impact of periodontitis on the progression of Alzheimer's disease: a prospective cohort study. Clin Oral Investig. 2023 Dec 30;28(1):67. doi: 10.1007/s00784-023-05445-w. PMID 38159159